CLINICAL TRIAL: NCT03367884
Title: Neck Dissection Versus Radiotherapy for Cervical Lymph Node Metastasis in Advanced Hypopharyngeal Carcinoma With Poor Response to Induction Chemotherapy : A Randomized Controlled Prospective Study
Brief Title: Neck Dissection vs Radiotherapy for Cervical Metastases in Advanced Hypopharyngeal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Tianjin Medical University Second Hospital (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJHPC-01
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Hypopharyngeal Carcinoma
Keywords: Hypopharyngeal cancer; Neck dissection; Induction chemotherapy; Cervical lymph node metastasis; definitive radiotherapy
MeSH Terms: conditions — Hypopharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck dissection group (Experimental): Neck dissection followed by radiotherapy(50Gy) according to risk factors
  Interventions: Procedure: Neck dissection followed by radiotherapy(50Gy) according to risk factors
- Radiotherapy group (Active Comparator): Definitive radiotherapy (70Gy)
  Interventions: Radiation: Definitive radiotherapy

INTERVENTIONS:
Procedure: Neck dissection followed by radiotherapy(50Gy) according to risk factors — Neck dissection followed by radiotherapy(50Gy) according to risk factors
  Arms: Neck dissection group
Radiation: Definitive radiotherapy — Definitive radiotherapy (70Gy)
  Arms: Radiotherapy group

SUMMARY:
At the time of diagnosis, approximately 60%-80% of patients with hypopharyngeal cancer are found with cervical lymph node metastasis. Cervical nodal metastasis is an important prognostic factor in hypopharyngeal cancer. Induction chemotherapy is frequently used in advanced hypopharynx cancer. However, sometimes CR was obtained at the tumor's primary site but not in the palpable lymph nodes in the neck, the large cervical lymph node metastasis poorly responded to induction chemotherapy in a considerable percentage of patients. At present, patients with primary tumor achieved CR preferred to receive definitive radiotherapy no matter cervical lymph node metastasis SD or progression. But, radiotherapy was poor effective to the big cervical lymph node metastasis, because the inner of big cervical lymph node metastasis was hypoxic and necrosis. The investigators conducted a prospective, randomised trial to compare neck dissection with definitive radiotherapy for advanced hypopharyngeal cancer cervical lymph node metastasis with poor response to induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document
2. Age≥ 18 and≤ 75 years
3. Histological/ cytological/ Imaging examination proven hypopharyngeal squamous-cell carcinoma in preoperative assessment
4. Advanced hypopharyngeal cancer with metastatic cervical lymph node more than 2cm in diameter
5. EPOG≤1,KPS≥ 70
6. No contraindication of surgery and radiotherapy
7. No serious disease history of the heart, liver, kidney, lung and other important organs
8. Expected survival period≥ 12 months
9. Good compliance

Exclusion Criteria:

1. Inability to provide an informed consent
2. Other malignancy tumor history,(except for cured skin basal cell carcinoma and papillary thyroid carcinoma)
3. Serious cardiovascular, liver, respiratory, kidney and neurologic and psychiatric disease with clinical symptoms
4. The patient has received prior surgery or radiotherapy (except for biopsy)
5. The patient has received chemotherapy or immunotherapy
6. Pregnant or lactating women
7. Other disease requiring simultaneous surgery or radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Neck control rates | 2 years
  The percentage of patients without cervical lymph node metastasis

SECONDARY OUTCOMES:
Disease-free survival | 1 year
  The proportion of patients did not find clear evidence of recurrence or metastasis
Disease-free survival | 2 years
  The proportion of patients did not find clear evidence of recurrence or metastasis
Disease-free survival | 3 years
  The proportion of patients did not find clear evidence of recurrence or metastasis
Disease-free survival | 5 years
  The proportion of patients did not find clear evidence of recurrence or metastasis
Overall survival | 3 years
  The proportion of patients who survived
Overall survival | 5 years
  The proportion of patients who survived
Quality of life(QOL) QLQ-C30 | 1 year
  Evaluated by the European Organization for Research and Treatment of Cancer(EORTC)QLQ-C30
Quality of life(QOL) QLQ-HN35 | 1 year
  Evaluated by the European Organization for Research and Treatment of Cancer(EORTC) QLQ-HN35

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Wang, Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China